CLINICAL TRIAL: NCT02963220
Title: Cognitive-Behavioral Therapy for Avoidant/Restrictive Eating Disorder: A Treatment Development and Pilot Study
Brief Title: Cognitive-Behavioral Therapy for Avoidant/Restrictive Food Intake Disorder: A Treatment Development and Pilot Study
Acronym: CBT-AR Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Psychological Foundation (Other); The Hilda & Preston Davis Foundation (Other)
Responsible Party: Principal Investigator, Jennifer Thomas, Co-Director, Eating Disorders Clinical and Research Program; Associate Professor of Psychology (Psychiatry), Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002108
Record Dates: First submitted 2016-10-31; First posted 2016-11-15 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Avoidant/Restrictive Food Intake Disorder (ARFID)
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CBT-AR (Experimental): There is only one arm in this study - all participants will be in the same arm, as all participants will receive CBT-AR. There is no control group.
  Interventions: Behavioral: CBT-AR

INTERVENTIONS:
Behavioral: CBT-AR — 20-30 sessions of cognitive behavioral therapy for avoidant/restrictive food intake disorder (CBT-AR), held once per week in an outpatient setting

SUMMARY:
The primary aim of this study is to pilot cognitive behavioral therapy (CBT-AR)for avoidant/restrictive food intake disorder (ARFID) in one study for children and adolescents (ages 10-17 years) and one study for adults (ages 18-65 years).

DETAILED DESCRIPTION:
This study is designed to pilot the CBT-AR treatment in youth with ARFID to determine treatment acceptability and efficacy.This includes evaluating the efficacy and acceptability of CBT-AR in reducing primary ARFID symptoms from pre- to post-treatment, and to assess whether improvement in individual symptoms is related to the timing of relevant interventions. The investigators hypothesize that from pre-treatment to post-treatment, subjects with ARFID will decrease severity of self-reported ARFID symptoms, decrease self-reported anxiety and depression, and improve psychosocial functioning. The investigators further hypothesize that overall, subjects with ARFID will have reduced phobic avoidance, sensory sensitivity, and/or low appetite in comparison to their pre-treatment symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Males and females; ages 10-17 years AND 18-65 years with avoidant/restrictive eating disorder or avoidant/restrictive eating patterns, characterized by either (i) Eating Disorder Assessment-5 (EDA-5) (ii) Kiddie Schedule for Affective Disorders and Schizophrenia for School Age Children-Present and Lifetime Version (KSADS-PL)

Exclusion Criteria:

* Use of systemic hormones, pregnancy or breastfeeding within eight weeks
* History of psychosis by KSADS-PL
* Substance or Alcohol Use Disorder active within the past month by KSADS-PL
* Active suicidal ideation
* Gastrointestinal tract surgery (including gastrectomy, gastric bypass surgery, and small or large bowel resection)
* Any feeding or eating disorder other than ARFID determined by EDA-5
* Any clinically significant disordered eating as evidenced by EDE-Q global > 4.0 or self-induced vomiting, laxatives, diuretics, purposeful fasting, or compensatory exercise in past 28 days
* Medical history of intellectual disability (IQ< 70)
* Has previously received more than 4 hours of CBT for ARFID in the past
* Is currently receiving another form of psychosocial treatment for ARFID (e.g., occupational therapy, speech therapy, another form of psychotherapy) and is unable to discontinue that treatment for the duration of this study.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-10; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Pica, ARFID, Rumination Disorder Interview (PARDI) severity score | Change from pre-treatment to after 20 weeks of CBT-AR (or 40 weeks, if the patient is underweight [BMI < 18.5 kg/m^2])
  A semi-structured interview to assess pica, ARFID, and/or rumination disorder diagnosis, severity, and symptoms

SECONDARY OUTCOMES:
BMI (kg/m^2) | Change from pre-treatment to after 20 weeks of CBT-AR (or 40 weeks, if the patient is underweight [BMI < 18.5 kg/m^2])
  If the patient is underweight, BMI will be used as an outcome measure
Food Neophobia Scale | Change from pre-treatment to after 20 weeks of CBT-AR (or 40 weeks, if the patient is underweight [BMI < 18.5 kg/m^2])
  Patient will complete the FNS prior to treatment and again after 20 (or 40 week) to assess change in reluctance to new foods
Parent PARDI | Change from pre-treatment to after 20 weeks of CBT-AR (or 40 weeks, if the patient is underweight [BMI < 18.5 kg/m^2])
  A semi-structured interview to assess pica, ARFID, and/or rumination disorder diagnosis, severity, and symptoms (based on parent report)
Child Depression Inventory 2 (CDI 2) score | Change from pre-treatment to after 20 weeks of CBT-AR (or 40 weeks, if the patient is underweight [BMI < 18.5 kg/m^2])
  Patient will complete the CDI 2 prior to treatment and again after 20 (or 40 weeks) to assess change in severity of depression
State-Trait Anxiety Inventory (STAI) score | Change from pre-treatment to after 20 weeks of CBT-AR (or 40 weeks, if the patient is underweight [BMI < 18.5 kg/m^2])
  Patient will complete the STAI prior to treatment and again after 20 (or 40 weeks) to assess change in severity of anxiety
Clinical Impairment Assessment (CIA) score | Change from pre-treatment to after 20 weeks of CBT-AR (or 40 weeks, if the patient is underweight [BMI < 18.5 kg/m^2])
  Patient will complete the CIA prior to treatment and again after 20 (or 40 weeks) to assess change in severity of clinical impairment
Hormone data | Change from pre-treatment to after 20 weeks of CBT-AR (or 40 weeks, if the patient is underweight [BMI < 18.5 kg/m^2])
  Patient will complete a test meal and we will collect blood at T0, T30, T60, and T120 prior to treatment and again after 20 (or 40) weeks of CBT-AR, in order to assess the change in hormone levels.
Functional magnetic resonance imaging (fMRI) | Change from pre-treatment to after 20 weeks of CBT-AR (or 40 weeks, if the patient is underweight [BMI < 18.5 kg/m^2])
  Patient will complete fMRI scan prior to treatment and again after 20 (or 40) weeks of CBT-AR, in order to assess the change in fMRI paradigms.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Thomas, Ph.D., Principal Investigator — Massachusetts General Hospital; Kamryn T. Eddy, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Eating Disorders Clinical and Research Program (Massachusetts General Hospital), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas JJ, Becker KR, Breithaupt L, Murray HB, Jo JH, Kuhnle MC, Dreier MJ, Harshman S, Kahn DL, Hauser K, Slattery M, Misra M, Lawson EA, Eddy KT. Cognitive-behavioral therapy for adults with avoidant/restrictive food intake disorder. J Behav Cogn Ther. 2021 Mar;31(1):47-55. doi: 10.1016/j.jbct.2020.10.004. Epub 2021 Mar 3. PMID 34423319